CLINICAL TRIAL: NCT04251923
Title: Vaginal Prolapse Surgery Accompanied by Mid Urethral Sling Versus no Sling for Reduction of Postoperative Incontinence: a Randomized Controlled Trial
Brief Title: Vaginal Prolapse Surgery Accompanied by Mid Urethral Sling Versus no Sling for Reduction of Postoperative Incontinence
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: B.P. Koirala Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, Baburam Dixit Thapa, Assistant Professor, Obstetrics and Gynecology, B.P. Koirala Institute of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRC/1536/019
Record Dates: First submitted 2020-01-15; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Stress Urinary Incontinence; Vaginal Hysterectomy; Quality of Life
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Hysterectomy, Vaginal

STUDY DESIGN:
Intervention Model Description: If patient gives consent and falls on selection criteria (inclusion and exclusion), she will be enrolled for randomization. Written informed consent will be taken. Computer generated simple randomization will be done.filled. POP-Q, Occult SUI and ESST will be checked and noted. This will be done by one of the researcher. Surgery will be performed by one of the researcher. Both Group I and Group II patients will undergo vaginal hysterectomy with McCall's culdoplasty and anterior repair with or without posterior repair according to the need. Patient who falls in Group I will undergo midurethral sling with tension free vaginal tape (TVT).
  Patient will be followed up at 3 and 6 months. The primary outcome of the study will be the difference in SUI. Secondary outcomes will be BFLUTS AND udi-6 SCORE, voiding dysfunction, dyspareunia, patient satisfaction and complications during surgery.
Who Masked: Outcomes Assessor
Masking Description: those who will be filling questionnaires before and after the surgery are masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- vagianl prolapse surgery accompanied with TVT sling (Experimental): patients will undergo vaginal hysterectomy with McCall's culdoplasty and anterior repair with or without posterior repair according to the need. Patient who falls in Group will undergo mid urethral sling with tension free vaginal tape (TVT) using TVT mid urethral sling.
  Interventions: Device: Retro pubic sling
- vaginal prolapse surgery not accompanied with sling (No Intervention): patients will undergo vaginal hysterectomy with McCall's culdoplasty and anterior repair with or without posterior repair according to the need.

INTERVENTIONS:
Device: Retro pubic sling — patient after hysterectomy will undergo retropubic sling surgery in the same setting. Retropubic sling will be inserted vaginally in the retropubic area following standard protocol.
  Other Names: vaginal hysterectomy
  Arms: vagianl prolapse surgery accompanied with TVT sling

SUMMARY:
Prevalence of pelvic organ prolapsed is high in Nepal. After prolapse surgery many patients are affected with incontinence. Incontinence has physical, social and mental effect to the individual. This study is designed to know the role for mid urethral sling during vaginal prolapse surgery to decrease the rate of incontinence after the surgery.

DETAILED DESCRIPTION:
Aim: To de termine the effect of mid urethral sling in reducing postoperative incontinence after vaginal prolapse surgery.

General Objectives: To compare the risk of de novo postoperative incontinence between prolapsed surgery with mid urethral sling versus no sling.

Specific Objectives: to compare the change in score of BFLUTS-SF (Bristol Female lower urinary tract symptoms- sexual function) and UDI-6 (Urinary distress inventory-6) pre and post surgery between the two groups.

Research Hypothesis: The use of mid urethral sling after vaginal prolapse surgery has role in reduction of postoperative incontinence.

Materials & Methods:

1. Whether study involves humans/animals or both : Humans
2. Population/ participants: Patients with pelvic organ prolapse who are planned for vaginal prolapse surgery in BPKIHS (BP Koirala Institute of Health and Sciences).
3. Type of study design: a randomized controlled trial

(e) Expected sample size: 54 Sample size calculation: Previous study done by Control groups: Patient undergoing vaginal prolapse surgery only without mid urethral sling. There will be small incision in the suprapubic region that mimics the TVT incision.

(f) Probable duration of study: one and half year (g) Setting: BPKIHS, Department of Obstetrics and Gynecology (h) Parameter/Variables to be applied/ measured: Age, BMI, POPQ (Pelvic organ prolapse quantification) stage, menopause, ESST (Empty supine stress test).

(i) Outcome measures: LUTS score, UDI-6 score, SUI (stress urinary incontinence), Voiding dysfunction, dyspareunia, satisfaction, Complications like bladder injury, hemorrhage.

(j) Rationale for statistical methods to be employed: attached (k) Ethical clearance: Study will be started after getting clearance from the IRC (Institutional review committee) of BPKIHS .

(l) Permission to use copyright questionnaire/Proforma: Pre designed Proforma and questionnaire will be used to collect the data. The internationally valid questionnaire in English will be validated in Nepali language first and then it will be used.

(m) Maintain the confidentiality of subject: The confidentiality of the patients will be maintained throughout the research.

ELIGIBILITY:
Inclusion Criteria:

* Clinical POP-Q stage 3 or more
* Must have cell phone

Exclusion Criteria:

* Patient with POPQ stage less than stage 3
* Patient not giving consent
* Patient with previous pelvic and spine surgery
* Patient having positive cough stress test on examination

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — all female patients
Enrollment: 56 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Stress urinary incontinence | 3 months
  The primary outcome of the study will be the presence of stress urinary incontinence in post operative at 3 months follow up. During follow up patient will be asked about the urinary incontinence on coughing, sneezing, heavy work and will examined in comfortably full bladder and cough stress test will be done to confirm the diagnosis of stress urinary incontinence.
stress urinary incontinence | 6 months
  The primary outcome of the study will be the presence of stress urinary incontinence in post operative at 6 months follow up. During follow up patient will be asked about the urinary incontinence on coughing, sneezing, heavy work and will examined in comfortably full bladder and cough stress test will be done to confirm the diagnosis of stress urinary incontinence.

SECONDARY OUTCOMES:
1) BFLUTS-FS (frequency symptoms), VS(voiding symptoms), IS (Irritable symptoms), Sex symptoms , QoL (Quality of life) score 2) UDI-6 (Urinary distress inventory-6) score 3) Complications during surgery 4) Dyspareunia 5) Pelvic pain | 3 months
  The main two questionnaires used in this study are BFLUTS-SF and UDI-6. BFLUTS-SF has five different section
  1. BFLUTS- FS: frequency symptoms and score ranges from 0-15, VS: voiding symptoms and score is from 0-12 IS: irritable bladder symptoms and score is from 0-20. . sex: sexual symptoms and score is from 0-6. QoL: quality of life due to bladder symptoms and score is from 0-18.
  2. UDI-6 score: quality of life due to bladder symptoms. Score range from 0-18. Severity increases as score increases in each section. High score denotes patient are highly affected due to bladder problems.
  3. Complications are noted hemorrhage, bladder injury, prolonged catheterization, urinary retention, need of mesh removal Remote complications: mesh erosion, Dyspareunia, pelvic pain, these complications will be noted. For pelvic pain visual analogue scale will be used, score having 1-10; 0, being least to 10 being the maximum.
1) BFLUTS-FS (frequency symptoms), VS(voiding symptoms), IS (Irritable symptoms), Sex symptoms , QoL (Quality of life) score 2) UDI-6 (Urinary distress inventory-6) score 3) Complications during surgery 4) Dyspareunia 5) Pelvic pain | 6 months
  The main two questionnaires used in this study are BFLUTS-SF and UDI-6. BFLUTS-SF has five different section
  1. BFLUTS- FS: frequency symptoms and score ranges from 0-15, VS: voiding symptoms and score is from 0-12 IS: irritable bladder symptoms and score is from 0-20. . sex: sexual symptoms and score is from 0-6. QoL: quality of life due to bladder symptoms and score is from 0-18.
  2. UDI-6 score: quality of life due to bladder symptoms. Score range from 0-18. Severity increases as score increases in each section. High score denotes patient are highly affected due to bladder problems.
  3. Complications are noted hemorrhage, bladder injury, prolonged catheterization, urinary retention, need of mesh removal Remote complications: mesh erosion, Dyspareunia, pelvic pain, these complications will be noted. For pelvic pain visual analogue scale will be used, score having 1-10; 0, being least to 10 being the maximum.

CONTACTS AND LOCATIONS:
Overall Officials: Mohan ch Regmi, Professor, Study Chair — BPKIHS

IPD SHARING:
Plan to Share IPD: No